CLINICAL TRIAL: NCT03780907
Title: A Randomised, Double-Blind, Placebo-Controlled Study of the Tolerability, Safety and Pharmacokinetics of E2007 in Epileptic Patients With Partial and Generalised Seizures
Brief Title: Safety and Pharmacokinetics Study of E2007 to Treat Partial and Generalised Seizures in People With Epilepsy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E2007-E049-203
Record Dates: First submitted 2015-07-31; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2015-11

CONDITIONS: Epilepsy
Keywords: Epilepsy; E2007; partial seizures; generalized seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — perampanel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- E2007 1 mg (Experimental): Tablet, once daily to be taken in the morning by mouth, one hour before breakfast, with a glass of water.
  Interventions: Drug: E2007
- E2007 2 mg (Experimental): Tablet, once daily to be taken in the morning by mouth, one hour before breakfast, with a glass of water.
  Interventions: Drug: E2007
- Placebo (Placebo Comparator): Tablet, once daily to be taken in the morning, one hour before breakfast, with a glass of water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: E2007 — 1 mg of E2007 was administered by mouth once daily.
  Arms: E2007 1 mg
Drug: E2007 — 2 mg of E2007 was administered by mouth once daily.
  Arms: E2007 2 mg
Drug: Placebo — Placebo once daily of oral tablet formulation to be taken in the morning, one hour before breakfast, with a glass of water.
  Arms: Placebo

SUMMARY:
The objectives of this study were to assess the tolerability and safety of E2007 in patients with refractory partial or generalised seizures and to assess the pharmacokinetics of E2007 in epileptic patients receiving at least one concomitant anti-epileptic drug.

ELIGIBILITY:
Inclusion Criteria

A patient who met the following inclusion criteria was eligible to participate in the study:

1. Males or females with simple or complex partial seizures with or without secondary generalization, or primary generalized tonic-clonic seizures according to the International League against Epilepsy classification. Patient records were to document the frequency of seizure.
2. Age: 18 to 65 years.
3. Race: any.
4. Patients receiving up to two additional anti-epileptic medications at doses that were stable for at least the four weeks immediately preceding baseline.
5. Patients willing and able to co-operate with the study procedures including completion of patient diaries.
6. Patients living at home with a partner or carer able to monitor compliance.
7. Patients giving informed consent to participate in the study.

Exclusion Criteria

A patient who met the following exclusion criteria was not eligible to participate in the study:

1. Pregnant or lactating women.
2. Women of childbearing potential unless (1) surgically sterile or (2) practicing effective contraception (eg, abstinence, IUD or barrier method plus hormonal method) and having a negative serum beta-HCG result at screening and being willing to remain on the current form of contraception for the duration of the study. Postmenopausal women could be included but were to have been amenorrhoeic for at least 12 months to be considered as not being of child-bearing potential.
3. Fertile men not willing to use reliable contraception or with partners not willing to use reliable contraception.
4. Patients with status epilepticus within the past 24 months.
5. Patients with unstable abnormalities of the hepatic, renal, cardiovascular, respiratory, abdominal, haematological, endocrine or metabolic systems which might complicate assessment of the tolerability of the study medication.
6. Patients with significantly elevated liver enzymes (abnormal bilirubin level, or serum transaminase levels more than 1.5 times the upper limit of normal).
7. Patients taking drugs other than anti-epileptic agents which induce the enzyme cytochrome P450 3A4 (since these might reduce the plasma concentration of E2007), including dexamethasone, rifabutin, rifampacin, St John's Wort.
8. Patients with past or present drug or alcohol abuse.
9. Patients with unstable psychiatric illness.
10. Patients who had received an investigational drug within the three months before baseline.
11. Patients without a reliable partner or carer.
12. Patients with any condition which would make the patient, in the opinion of the investigator, unsuitable for the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2003-02-14 (Actual); Primary Completion 2003-08-06 (Actual); Study Completion 2003-08-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAEs) | From administration of first dose of study drug up until 42 days.
  The TEAEs were defined as those Adverse Events (AEs) that start on or after the first dose of the treatment until the end of the study. AEs were classified by the investigator as 'not related', 'possibly related' or 'probably related'.
Clinical Global Impression of Tolerability (CGIT) | Day 28
  The investigator's global impressions of the tolerability of the study treatment was based on a five point scale: 1 - very good, 2 - good, 3 - moderate, 4 - poor, and 5 - very poor.
Pharmacokinetic Parameter: Area Under the Curve (AUC)(0-24hr) of E2007 | Day 1 and Day 14
  Standard pharmacokinetic parameters for E2007 were derived from plasma drug concentrations in epileptic participants. A measure of systemic drug exposure over 24 hours, which is obtained by collecting a series of blood samples and measuring the concentrations of drug in each sample.
Pharmacokinetic Parameter: Cmax (Maximum Observed Plasma Concentration) of E2007 | Day 1 and Day 14
  Standard pharmacokinetic parameters for E2007 were derived from plasma drug concentrations in epileptic participants. The maximum concentration of a drug observed after its administration.
Pharmacokinetic Parameter: Tmax (Time to Maximum Concentration) of E2007 | Day 1 and Day 14
  Standard pharmacokinetic parameters for E2007 were derived from plasma drug concentrations in epileptic participants. The time after dosing when a drug attains its highest measurable concentration (Cmax).
Pharmacokinetic Parameter: Css,min (Minimum Steady State Plasma Concentration) of E2007 | Day 14
  Standard pharmacokinetic parameters for E2007 were derived from plasma drug concentrations in epileptic participants. Lowest plasma concentration within a steady-state dosing interval.
Pharmacokinetic Parameter: Cav (Average Plasma Concentration) of E2007 | Day 14
  Standard pharmacokinetic parameters for E2007 were derived from plasma drug concentrations in epileptic participants.
Pharmacokinetic Parameter: Peak-to-trough Fluctuation (PTF) of E2007 | Day 14
  Standard pharmacokinetic parameters for E2007 were derived from plasma drug concentrations in epileptic participants.
Pharmacokinetic Parameter: Observed Accumulation Ratio (Rac) of E2007 | Day 14
  Standard pharmacokinetic parameters for E2007 were derived from plasma drug concentrations in epileptic participants.

SECONDARY OUTCOMES:
Change from Baseline of Bond and Lader Scale | Baseline, Day 28 and Day 42
  The Bond and Lader visual analogue mood scale (VAMS) had a score from 0 - 100; a higher score represented worsening of the participants condition attributed to 3 factors, (1) Anxiety (e.g., calmness), (2) Sedation (e.g., alertness, (3) Dysphoria (e.g., contentedness). The change was visit minus baseline.
Change from Baseline of Peak Saccadic Velocity (PSV) | Baseline, Day 28, Day 42
  Saccadic velocity is the rate of eye movement in response to stimulus. The saccadic eye movement was used to allow comparison of any sedative effects seen.
Number of Particpants receiving other Anti-epileptic agents During Treatment | Day 1 and Day 14
Percent Change from Baseline of Failed Saccades | Baseline, Day 28, Day 42
  Failed saccades is stimulus resulting in no eye movement above a defined threshold within a specified time.
Mean trough concentrations of E2007 | Day 7, Day 21, and Day 28
Number of seizures | Baseline (Day-1) to Day 42
The Clinical Global Impression of Change | Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- 3ClinicalResearch AG, Hennigsdorf, Germany

REFERENCES:
- [Derived] Maguire M. Response to "Perampanel and pregnancy: Could experience be a gloomy lantern that does not even illuminate its bearer?". Epilepsy Behav. 2022 Apr;129:108654. doi: 10.1016/j.yebeh.2022.108654. Epub 2022 Mar 16. No abstract available. PMID 35305920